CLINICAL TRIAL: NCT02144948
Title: Pilot Study to Investigate the Effect of E-coli-nissle as Probiotic Adjuvant to Antidiabetic Standard Care in Patients With Diabetes Mellitus Type II
Brief Title: Investigation of the Effect of E.-Coli-Nissle as Supporting Therapy to Standard Care of Diabetes Mellitus Type II
Acronym: PUNiDIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Ardeypharm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUNiDIA-2014
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2015-08

CONDITIONS: Diabetes Mellitus Type II
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E.-coli-Nissle (Experimental): 10 patients will be enrolled Intervention: E.-coli-Nissle (Mutaflor), oral suspension Dose: 1 ml / day frequency: qd
  Interventions: Drug: e.-coli-nissle

INTERVENTIONS:
Drug: e.-coli-nissle — 1 ml qd for 24 weeks
  Other Names: Mutaflor

SUMMARY:
This is a pilot study to investigate the effect of e.-coli-nissle as supporting therapy to antidiabetic standard care in patients with diabetes mellitus type II

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus type 2;
* HbA1c >7 % (stable für 6 months, max. variation of 0,5%)
* stable oral antidiabetic therapy for 6 months with Metformin, Vildagliptin, Gliniden or without oral Antidiabetics
* age of 45 to <80 years (men and women)

Exclusion Criteria:

* Myocardial infarction or stroke within the last 5 years
* Therapy with acarbose
* Acute peripheral arterial disease within the last 12 months
* Instable metabolic situation
* Uncontrolled hypertension
* Body-Mass-Index ≥ 35 kg/m²
* Smokers
* Daily consumption of probiotic food
* Malignant disease within the last 5 years
* Status post transplantation
* Immunosuppressive therapy within the last 3 months
* Therapy with antibiotics
* Macroalbuminuria
* Severe liver disease

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Decrease in HbA1c levels | 24 weeks

SECONDARY OUTCOMES:
change in insulin resistance/secretion | 24 weeks
change in lipid parameters | 24 weeks
change in parameters of oxidative stress | 24 weeks
change in gastrointestinal condition | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antje Bergmann, Prof.Dr.med., Principal Investigator — Carus Hausarztpraxis on behalf of GWT-TUD GmbH; Stefan R. Bornstein, Prof.Dr.med, Study Chair — Universitätsklinikum Dresden on behalf of GWT-TUD GmbH
Locations (1):
- Carus-Hausarztpraxis, Dresden, Germany